CLINICAL TRIAL: NCT02938858
Title: The French Registry on the First-line Treatment of Non High-risk Acute Promyelocytic Leukemia (APL) in Patients Aged ≤ 70 Years
Brief Title: French Registry of First-line Treatment of Acute Promyelocytic Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: French registry APL
Record Dates: First submitted 2016-09-22; First posted 2016-10-19 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ATRA-chimio: according to usual practice center
- ATRA-ATO: according to usual practice center

SUMMARY:
The registry aims to compare the two first-line available treatment approaches in non-high-risk APL patients aged ≤ 70 years - ATRA plus chemotherapy and ATRA plus ATO - in terms of practitioner's choice between the two options, clinical effectiveness and cost-effectiveness, long-term outcome, and short- and long-term toxic effects.

DETAILED DESCRIPTION:
* Collection of epidemiological data on non-high-risk APL patients aged ≤ 70 years: age and sex distribution, medical history, prognostic factors (time to treatment start, severity of coagulopathy at presentation, Performance status…).
* Documentation of clinical and biologic effectiveness of the two first-line treatment approaches available for non-high-risk APL patients.
* Documentation of Minimal Residual Disease (MRD).
* Correlation of clinical outcomes with the chosen therapy.
* Validation of published prognostic factors and identification of new prognostic factors

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed APL (either de novo or therapy-related) based on cytologic criteria and confirmed by the presence of the t(15;17) translocation and/or by the detection of the fusion transcript PML/RARα.
* Non-high-risk APL (White Blood Count < 10000/μl at presentation)
* Age ≤ 70 years

Exclusion Criteria:

* Relapsed APL
* Newly-diagnosed High-risk APL (White Blood Count > 10000/μl at presentation)
* Age > 70 years

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French patients with newly-diagnosed de novo or therapy-related non-high-risk APL (White Blood Count < 10000/μl) aged ≤ 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | From date of induction until the date of first documented event, assessed up to 60 months
  events are: no achievement of haematological complete remission after induction therapy; no achievement of molecular remission after the consolidation courses; relapse; death including early death

SECONDARY OUTCOMES:
Rate of hematological complete remission | up to 30 days
  from date of inclusion until end of induction therapy
Rate of overall survival | at 5 years
  Overall survival defined as the time from inclusion until death or end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FENAUX, MD, Principal Investigator — French APL Cooperative Group
Locations (27):
- France (27):
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - Groupe Hospitalier SUD, Amiens
  - Centre Hospitalier V. Dupouy, Argenteuil
  - Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux Pellegrin enfant, Bordeaux
  - CHRU de Brest - Pédiatrie Spécialisée, Brest
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hopital Andre Mignot, Le Chesnay
  - CH Dr Schaffner, Lens
  - Chru - Hopital Claude Huriez, Lille
  - Hôpital universitaire Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - Chu Timone, Marseille
  - CHR Metz-Thionville - Hôpital de Marcy, Metz
  - CHU Saint Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital de la Source, Orléans
  - Hôpital TROUSSEAU, Paris
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris
  - CHU Hôpital Sud - service Hémato-oncologie Pédiatrique, Rennes
  - Hôpital V. Provo, Roubaix
  - Centre Henri Becquerel, Rouen
  - Institut de Cancerologie de La Loire, Saint-Priest-en-Jarez
  - IUCT Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No